CLINICAL TRIAL: NCT00883337
Title: A Multi-center, Randomized, Parallel-group, Rater-blinded Study Comparing the Effectiveness and Safety of Teriflunomide and Interferon Beta-1a in Patients With Relapsing Multiple Sclerosis Plus a Long Term Extension Period
Brief Title: A Study Comparing the Effectiveness and Safety of Teriflunomide and Interferon Beta-1a in Patients With Relapsing Multiple Sclerosis
Acronym: TENERE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EFC10891; 2008-006226-34 (EudraCT Number)
Record Dates: First submitted 2009-04-16; First posted 2009-04-17 (Estimated); Results first posted 2012-11-06 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-05

CONDITIONS: Multiple Sclerosis
Keywords: Relapsing-remitting multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting | interventions — Interferon beta-1a; teriflunomide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Teriflunomide 7 mg / 14 mg (Experimental): Teriflunomide 7 mg once daily (core treatment period) and teriflunomide 14 mg once daily (extended treatment period).
  Interventions: Drug: Teriflunomide
- Teriflunomide 14 mg / 14 mg (Experimental): Teriflunomide 14 mg once daily (core treatment period) and teriflunomide 14 mg once daily (extension treatment period).
  Interventions: Drug: Teriflunomide
- IFN-β-1a / 14 mg (Active Comparator): Interferon β-1a 3 times a week (core treatment period) and teriflunomide 14 mg once daily (extended treatment period).
  Interventions: Drug: Interferon β-1a; Drug: Teriflunomide

INTERVENTIONS:
Drug: Interferon β-1a — Sterile preservative-free solution packaged in graduated pre-filled syringes
  Subcutaneous injection
  Ascending doses from 8.8 to 44 mcg according to local standard for Rebif®
  Other Names: Rebif®
  Arms: IFN-β-1a / 14 mg
Drug: Teriflunomide — Film-coated tablet
  Oral administration
  Other Names: HMR1726

SUMMARY:
Primary objective was to assess the effectiveness evaluated by the time to failure of two doses of teriflunomide in comparison to interferon beta-1a in participants with relapsing Multiple Sclerosis [MS].

Secondary objectives were:

* To assess the effect of the two doses in comparison to interferon beta-1a on:

  * Frequency of relapses,
  * Fatigue,
  * Participant's satisfaction with treatment.
* To evaluate the safety and tolerability of the two doses in comparison to interferon beta-1a.

The study consisted of a core treatment period with a common end date defined as 48 weeks after randomization of the last participant, followed by an optional long-term extension treatment period until teriflunomide is commercially available in accordance with local regulations.

DETAILED DESCRIPTION:
The core treatment period per participant was variable depending on the enrollment in the study (maximum of approximatively 118 weeks). The two doses of teriflunomide were administered in double-blind fashion, whereas interferon beta-1a (Rebif®) was open-label.

The opportunity to continue with the highest dose of teriflunomide in open-label fashion was offered to the participants who successfully completed treatment in the core study.

The overall treatment period was followed by a 4-week elimination follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing form of MS meeting McDonald's criteria for MS diagnosis and Expanded Disability Status Scale [EDSS] score ≤5.5 at screening visit.

Exclusion Criteria:

* Significantly impaired bone marrow function or, significant anemia, leukopenia or thrombocytopenia;
* Persistent significant or severe infection.
* Liver function impairment or known history of hepatitis.
* Use of adrenocorticotrophic hormone [ACTH] or systemic corticosteroids for 2 weeks prior to randomization.
* Human immunodeficiency virus [HIV] positive.
* Prior use of Rebif®, or prior or concomitant use of other interferons in the 3 months prior to randomization.
* Prior or concomitant use of cladribine, mitoxantrone, or other immunosuppressant agents such as azathioprine, cyclophosphamide, cyclosporin, methotrexate, mycophenolate, or natalizumab.
* Pregnant or breast-feeding woman.

Extension criteria:

The participants who met all the following criteria at the end of the core study period were eligible for enrolment into the open-label extension phase:

* Participants who had not discontinued treatment in the core period and who had a minimum treatment of 48 weeks and completed the EOT visit (Visit 18).
* Participants who had not met criteria for treatment withdrawal.
* An informed consent must be obtained in writing from the participant for this open-label extension phase prior to entering and prior to completion of any extension phase procedure.
* Participants who demonstrated a willingness and ability to roll over to the extension phase with the opportunity to continue treatment on 14 mg/day of teriflunomide under open-label.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2009-04; Primary Completion 2011-09 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (54):
- Belgium (3):
  - Investigational Site Number 056003, Brussels
  - Investigational Site Number 056001, Ghent
  - Investigational Site Number 056002, Hasselt
- Canada (3):
  - Investigational Site Number 124003, Lévis
  - Investigational Site Number 124002, London
  - Investigational Site Number 124004, St. John's
- Czechia (3):
  - Investigational Site Number 203004, Jihlava
  - Investigational Site Number 203003, Prague
  - Investigational Site Number 203002, Prague
- France (5):
  - Investigational Site Number 250003, Bordeaux
  - Investigational Site Number 250005, Clermont-Ferrand
  - Investigational Site Number 250004, Lille
  - Investigational Site Number 250001, Montpellier
  - Investigational Site Number 250002, Strasbourg
- Germany (11):
  - Investigational Site Number 276003, Bad Mergentheim
  - Investigational Site Number 276011, Berlin
  - Investigational Site Number 276012, Berlin
  - Investigational Site Number 276001, Bochum
  - Investigational Site Number 276005, Dresden
  - Investigational Site Number 276007, Erbach im Odenwald
  - Investigational Site Number 276006, Essen
  - Investigational Site Number 276004, Halle
  - Investigational Site Number 276010, Hanover
  - Investigational Site Number 276009, Mainz
  - Investigational Site Number 276002, Münster
- Greece (2):
  - Investigational Site Number 300001, Athens
  - Investigational Site Number 300002, Thessaloniki
- Hungary (6):
  - Investigational Site Number 348001, Budapest
  - Investigational Site Number 348005, Budapest
  - Investigational Site Number 348003, Budapest
  - Investigational Site Number 348002, Esztergom
  - Investigational Site Number 348007, Kecskemét
  - Investigational Site Number 348004, Veszprém
- Italy (9):
  - Investigational Site Number 380010, Ancona
  - Investigational Site Number 380005, Bari
  - Investigational Site Number 380008, Cagliari
  - Investigational Site Number 380003, Cefalù
  - Investigational Site Number 380007, Genova
  - Investigational Site Number 380001, Milan
  - Investigational Site Number 380004, Pavia
  - Investigational Site Number 380002, Roma
  - Investigational Site Number 380006, Torino
- Poland (4):
  - Investigational Site Number 616002, Bialystok
  - Investigational Site Number 616004, Gdansk
  - Investigational Site Number 616003, Lublin
  - Investigational Site Number 616001, Warsaw
- Spain (4):
  - Investigational Site Number 724007, Barcelona
  - Investigational Site Number 724001, Bilbao
  - Investigational Site Number 724002, Majadahonda
  - Investigational Site Number 724003, Murcia
- Investigational Site Number 756002, Sankt Gallen, Switzerland
- Investigational Site Number 788002, Monastir, Tunisia
- United Kingdom (2):
  - Investigational Site Number 826002, London
  - Investigational Site Number 826003, Plymouth

REFERENCES:
- [Result] Vermersch P, Czlonkowska A, Grimaldi LM, Confavreux C, Comi G, Kappos L, Olsson TP, Benamor M, Bauer D, Truffinet P, Church M, Miller AE, Wolinsky JS, Freedman MS, O'Connor P; TENERE Trial Group. Teriflunomide versus subcutaneous interferon beta-1a in patients with relapsing multiple sclerosis: a randomised, controlled phase 3 trial. Mult Scler. 2014 May;20(6):705-16. doi: 10.1177/1352458513507821. Epub 2013 Oct 14. PMID 24126064
- [Derived] Comi G, Freedman MS, Meca-Lallana JE, Vermersch P, Kim BJ, Parajeles A, Edwards KR, Gold R, Korideck H, Chavin J, Poole EM, Coyle PK. Prior treatment status: impact on the efficacy and safety of teriflunomide in multiple sclerosis. BMC Neurol. 2020 Oct 6;20(1):364. doi: 10.1186/s12883-020-01937-4. PMID 33023488

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment initiated in April 2009 was completed in July 2010. A total of 369 participants were screened at 54 sites in 13 countries.
  The common end date of core treatment period was 14 September 2011 (maximum treatment duration of 115 weeks).
  The end date of extension was 13 May 2015 (maximum treatment duration of 197 weeks)
Pre-assignment Details: Randomization was stratified by country and baseline disability (Expanded Disability Status Scale [EDSS] score ≤3.5 or >3.5).
  Assignment to groups was done centrally using an Interactive Voice Response System (IVRS] in a 1:1:1 ratio after confirmation of the selection criteria. 324 participants were randomized at 53 sites.
Groups:
- Teriflunomide 7 mg/14 mg: Core treatment period: Teriflunomide 7 mg once daily.
  Extension treatment period: Teriflunomide 14 mg once daily.
- Teriflunomide 14 mg/14 mg: Core treatment period: Teriflunomide 14 mg once daily.
  Extension treatment period: Teriflunomide 14 mg once daily.
- IFN-β-1a / Teriflunomide 14 mg: Core treatment period: Interferon β-1a 3 times a week.
  Extension treatment period: Teriflunomide 14 mg once daily.
Period: Core Treatment Period
Arm/Group | Teriflunomide 7 mg/14 mg | Teriflunomide 14 mg/14 mg | IFN-β-1a / Teriflunomide 14 mg
Started | 109 | 111 | 104
Treated | 109 | 111 (One participant received teriflunomide 7 mg instead of teriflunomide 14 mg) | 101 (3 participants refused treatment with Rebif®)
Completed | 89 | 89 | 71
Not Completed | 20 | 22 | 33
Not completed — Adverse Event | 9 | 12 | 22
Not completed — Lack of Efficacy | 7 | 4 | 2
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 6
Not completed — Wish to be pregnant | 1 | 2 | 1
Not completed — Poor compliance to protocol | 0 | 0 | 1
Not completed — Other than above | 0 | 1 | 1
Period: Extension Treatment Period
Arm/Group | Teriflunomide 7 mg/14 mg | Teriflunomide 14 mg/14 mg | IFN-β-1a / Teriflunomide 14 mg
Started | 89 | 89 | 59 (12 participants completed the core period but didn't enter the extension period.)
Completed | 61 | 66 | 40
Not Completed | 28 | 23 | 19
Not completed — Adverse Event | 8 | 5 | 5
Not completed — Lack of Efficacy | 8 | 8 | 8
Not completed — Poor compliance to protocol | 1 | 1 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Other than above | 10 | 9 | 5

BASELINE CHARACTERISTICS:
Groups:
- Teriflunomide 7 mg / 14 mg: Core treatment period: Teriflunomide 7 mg once daily
  Extension treatment period: Teriflunomide 14 mg once daily
- IFNβ1a / Teriflunomide 14 mg: Core treatment period: Interferon β-1a 3 times a week.
  Extension treatment period: Teriflunomide 14 mg once daily.
- Total: Total of all reporting groups
Arm/Group | Teriflunomide 7 mg / 14 mg | Teriflunomide 14 mg/14 mg | IFNβ1a / Teriflunomide 14 mg | Total
Number analyzed (Participants) | 109 | 111 | 104 | 324
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.5 (9.2) | 36.8 (10.3) | 37.0 (10.6) | 36.3 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 78 | 71 | 219
  Male | 39 | 33 | 33 | 105
Region of enrollment [Number; unit: participants] — Due the small sample size in some countries, the countries were pooled as follows:
  * North America: Canada;
  * Eastern Europe: Czech Republic, Greece, Hungary and Poland;
  * Western Europe: Belgium, France, Germany, Italy, Spain, Switzerland and United Kingdon;
  '*' the only participant in Tunisia was included in the Western Europe group.
  participants
    North America | 8 | 6 | 7 | 21
    Eastern Europe | 39 | 41 | 35 | 115
    Western Europe* | 62 | 64 | 62 | 188
Time since first diagnosis of Multiple Sclerosis [MS] [Mean (Standard Deviation); unit: years] | 3.72 (5.19) | 3.68 (6.24) | 3.82 (5.69) | 3.74 (5.71)
Number of MS relapses [Median (Full Range); unit: relapses]
  Within the past year | 1 [0 to 3] | 1 [0 to 4] | 1 [0 to 5] | 1 [0 to 5]
  Within the past 2 years | 2 [0 to 4] | 2 [0 to 4] | 2 [0 to 6] | 2 [0 to 6]
Time since most recent MS relapse onset [Mean (Standard Deviation); unit: months] — The information was not available for one participant in the Teriflunomide 14 mg group
  months | 9.00 (13.96) | 7.90 (10.34) | 9.79 (10.72) | 8.88 (11.79)
MS subtype [Number; unit: participants]
  Relapsing Remitting | 109 | 108 | 104 | 321
  Secondary Progressive | 0 | 1 | 0 | 1
  Progressive Relapsing | 0 | 2 | 0 | 2
Baseline EDSS score [Number; unit: participants] — EDSS is an ordinal scale in half-point increments that qualifies disability in patients with MS. It consists of 8 ordinal rating scales assessing seven functional systems (visual, brainstem, pyramidal, cerebellar, sensory, bowel/bladder and cerebral) as well as ambulation.
  EDSS total score ranges from 0 (normal neurological examination) to 10 (death due to MS).
  participants
    ≤3.5 | 96 | 95 | 93 | 284
    >3.5 | 13 | 16 | 11 | 40

OUTCOME MEASURES:

1. Primary Outcome: Core Treatment Period: Overview of Failures
Description: Failure was defined as the first occurence of confirmed relapse or permanent treatment discontinuation (for any cause) which ever came first. If no events occurred, the participant was considered free of failure.
  Each episode of relapse - appearance, or worsening of a clinical symptom that was stable for at least 30 days, that persisted for a minimum of 24 hours in the absence of fever - was to be confirmed by an increase in Expanded Disability Status Scale [EDSS] score or Functional System scores.
Time Frame: Core treatment period between 48 and 118 weeks depending on when the participant was enrolled
Population: Intent-to-treat population: all randomized participants. Participants were considered in the treatment group to which they were randomized regardless of the drug they actually received.
Measure: Number; unit: participants
Groups:
- Teriflunomide 7 mg: Teriflunomide 7 mg once daily
- Teriflunomide 14 mg: Teriflunomide 14 mg once daily
- IFN-β-1a: Interferon β-1a 3 times a week
Arm/Group | Teriflunomide 7 mg | Teriflunomide 14 mg | IFN-β-1a
Number analyzed (Participants) | 109 | 111 | 104
participants
  Failure | 53 | 42 | 44
  Free of failure | 56 | 69 | 60

2. Primary Outcome: Core Treatment Period: Time to Failure: Kaplan-Meier Estimates of the Rate of Failure at Timepoints
Description: Probability of disability progression at 24, 48 and 96 weeks was estimated using Kaplan-Meier method on the time to failure defined as the time from randomization to failure. Participants free of failure were censored at the date of last treatment.
  Kaplan-Meier method consists in computing probabilities of non occurrence of event at any observed time of event and multiplying successive probabilities for time ≤t by any earlier computed probabilities to estimate the probability of being event-free for the amount of time t. Probability of event at time t is 1 minus the probability of being event-free for the amount of time t.
Time Frame: Core treatment period between 48 and 118 weeks depending on when the participant was enrolled
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | Teriflunomide 7 mg | Teriflunomide 14 mg | IFN-β-1a
Number analyzed (Participants) | 109 | 111 | 104
percent probability
  Probability of failure at 24 weeks | 25.7 [17.5 to 33.9] | 24.3 [16.3 to 32.3] | 29.8 [21.0 to 38.6]
  Probability of failure at 48 weeks | 35.8 [26.8 to 44.8] | 33.3 [24.6 to 42.1] | 36.5 [27.3 to 45.8]
  Probability of failure at 96 weeks | 58.8 [46.1 to 71.4] | 41.1 [30.9 to 51.4] | 44.4 [34.3 to 54.4]
Statistical Analysis 1: Comparison: Teriflunomide 14 mg vs IFN-β-1a; The study was sized to detect a difference between Teriflunomide and Rebif groups in the time to failure at a significance level of 0.025 with a power of 81%. Null hypothesis: * H1: No difference between Teriflunomide 14 mg and Rebif * H2: No difference between Teriflunomide 7 mg and Rebif; Test type: Superiority or Other; p = 0.5953, Log Rank — Hochberg testing procedure: * a-priori threshold for statistical significance ≤0.05 for the largest p-value of the 2 pair-wise comparisons * a-priori threshold for statistical significance ≤0.025 for the other p-value if the largest p-value >0.05; Two-sided Log Rank test with the region of enrollment and baseline EDSS stratum as stratification factors
Statistical Analysis 2: Comparison: Teriflunomide 7 mg vs IFN-β-1a; Null hypothesis: * H1: No difference between Teriflunomide 14 mg and Rebif * H2: No difference between Teriflunomide 7 mg and Rebif; Test type: Superiority or Other; p = 0.5190, Log Rank — [p-value comment as in outcome 2, analysis 1]; Two-sided Log Rank test with the region of enrollment and baseline EDSS stratum as stratification factors

3. Secondary Outcome: Core Treatment Period: Annualized Relapse Rate [ARR] - Poisson Regression Estimates
Description: ARR is obtained from the total number of confirmed relapses that occured during the treatment period divided by the sum of the treatment durations.
  To account for the different treatment durations among participants, a Poisson regression model with robust error variance was used (total number of confirmed relapses as response variable; log-transformed treatment duration as "offset" variable; treatment group, region of enrollment and baseline EDSS stratum as covariates).
Time Frame: Core treatment period between 48 and 118 weeks depending on when the participant was enrolled
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: relapses per year
Arm/Group | Teriflunomide 7 mg | Teriflunomide 14 mg | IFN-β-1a
Number analyzed (Participants) | 109 | 111 | 104
relapses per year | 0.410 [0.265 to 0.636] | 0.259 [0.153 to 0.438] | 0.216 [0.113 to 0.415]

4. Secondary Outcome: Core Treatment Period: Change From Baseline in Fatigue Impact Scale (FIS) Total Score
Description: FIS is a subject-reported scale that qualifies the impact of fatigue on daily life in patients with MS. It consists of 40 statements that measure fatigue in three areas; physical, cognitive, and social.
  FIS total score ranges from 0 (no problem) to 160 (extreme problem).
  Least-square means were estimated using a Mixed-effect model with repeated measures [MMRM] on FIS total score data (treatment group, region of enrollment, baseline EDSS stratum, visit, treatment-by-visit interaction, baseline value, and baseline-by-visit interaction as factors).
Time Frame: Baseline (before randomization) and 48 weeks
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Teriflunomide 7 mg | Teriflunomide 14 mg | IFN-β-1a
Number analyzed (Participants) | 109 | 111 | 104
units on a scale | 0.97 (2.96) | 4.10 (3.03) | 9.10 (3.21)

5. Secondary Outcome: Core Treatment Period: Treatment Satisfaction Questionnaire for Medication [TSQM] Scores
Description: TSQM version 1.4 is an instrument to assess patients' satisfaction with medication. It consists of 13 questions that cover three dimensions (effectiveness, side effects and convenience) plus a global satisfaction question. Four scores ranging from 0 to 100 (extremely satisfied) are obtained. Least-square means were estimated using a Mixed-effect model with repeated measures [MMRM] on TSQM score data (treatment group, region of enrollment, baseline EDSS stratum, visit, treatment-by-visit interaction as factors).
Time Frame: 48 weeks
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Teriflunomide 7 mg | Teriflunomide 14 mg | IFN-β-1a
Number analyzed (Participants) | 109 | 111 | 104
units on a scale
  Effectivness score | 67.25 (2.70) | 63.13 (2.75) | 59.30 (2.97)
  Side effects score | 95.29 (2.31) | 93.15 (2.34) | 71.38 (2.50)
  Convenience score | 88.30 (1.97) | 89.85 (1.98) | 61.90 (2.11)
  Global satisfaction score | 68.29 (2.77) | 68.82 (2.78) | 60.98 (2.94)

6. Secondary Outcome: Core Treatment Period: Overview of Adverse Events [AE]
Description: AE are any unfavorable and unintended sign, symptom, syndrome, or illness observed by the investigator or reported by the participant during the study.
Time Frame: from first study drug intake up to 112 days after last intake in the core treatment period or up to first intake in the extension treatment period, whichever occurred first
Population: Safety population: all randomized and treated participants. Participants were considered according to the drug actually received.
  The participant randomized to Teriflunomide 14 mg group who received Teriflunomide 7 mg was analyzed in the Teriflunomide 7 mg group.
Measure: Number; unit: participants
Arm/Group | Teriflunomide 7 mg | Teriflunomide 14 mg | IFN-β-1a
Number analyzed (Participants) | 110 | 110 | 101
participants
  Any AE | 103 | 102 | 97
  - Any serious AE | 12 | 6 | 7
  - Any AE leading to death | 0 | 0 | 0
  - Any AE leading to treatment discontinuation | 9 | 12 | 22

7. Secondary Outcome: Extension Treatment Period: Overview of AEs
Description: AEs were any unfavourable and unintended sign, symptom, syndrome, or illness observed by the investigator or reported by the participant during the study.
Time Frame: From first intake of study drug in extension treatment period up to 28 days after the last intake in the extension treatment period
Population: Safety population. Participants were considered in the treatment group to which they were randomized regardless of the drug they actually received.
Measure: Number; unit: participants
Groups:
- Teriflunomide 7 mg / 14 mg: Core treatment period: Teriflunomide 7 mg once daily. Extension treatment period: Teriflunomide 14 mg once daily.
- Teriflunomide 14 mg / 14 mg: Core treatment period: Teriflunomide 14 mg once daily. Extension treatment period: Teriflunomide 14 mg once daily.
- IFN-β-1a / 14 mg: Core treatment period: Interferon β1a 3 times a week. Extension treatment period: Teriflunomide 14 mg once daily.
Arm/Group | Teriflunomide 7 mg / 14 mg | Teriflunomide 14 mg / 14 mg | IFN-β-1a / 14 mg
Number analyzed (Participants) | 90 | 88 | 59
participants
  Any AE | 83 | 76 | 48
  Any serious AE | 9 | 13 | 12
  Any AE leading to death | 0 | 0 | 0
  Any AE leading to treatment discontinuation | 8 | 6 | 5

8. Secondary Outcome: Extension Treatment Period: ARR Poisson Regression Estimates
Description: ARR was obtained from the total number of confirmed relapses that occurred during the treatment period divided by the sum of the standardized treatment durations.To account for the different treatment durations among participants, a Poisson Regression Model with robust error variance was used (total number of confirmed relapses as response variable; log-transformed treatment duration as "offset" variable; treatment group, region of enrolment and baseline EDSS stratum as covariates).
Time Frame: Extension treatment period (Maximum: 197 weeks)
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: relapses per year
Arm/Group | Teriflunomide 7 mg / 14 mg | Teriflunomide 14 mg / 14 mg | IFN-β-1a / 14 mg
Number analyzed (Participants) | 89 | 89 | 59
relapses per year | 0.236 [0.154 to 0.362] | 0.193 [0.121 to 0.307] | 0.252 [0.145 to 0.438]

ADVERSE EVENTS:
Time Frame: AEs were collected from signature of the Informed Consent Form up to the last visit (197 weeks) in the study.
Description: The analysis was performed on the safety population as previously defined and included all AE that developed or worsened from first intake of study drug in extension treatment period up to 28 days after the last intake in the extension study treatment period.
Groups:
- Core Treatment Period: Teriflunomide 7 mg: Teriflunomide 7 mg once daily (mean exposure of 456.62 days).
- Core Treatment:Teriflunomide 14 mg: Teriflunomide 14 mg once daily (mean exposure of 434.43 days).
- Core Treatment: IFN-β-1a: Interferon β-1a 3 times a week (mean exposure of 405.18 days).
- Extended Treatment: Teriflunomide 14 mg (After 7 mg): Teriflunomide 14 mg once daily in extended treatment period after 7 mg in the core treatment period (mean exposure of 996.76 days).
- Extended Treatment: Teriflunomide 14 mg (After 14 mg): Teriflunomide 14 mg once daily in extended treatment period after 14 mg in core treatment period (mean exposure of 1015.32 days).
- Extended Treatment: Teriflunomide 14 mg (After IFN-β-1a): Teriflunomide 14 mg once daily in extended treatment period after Interferon β-1a 3 times a week in core treatment period (mean exposure of 1000.03 days).
Arm/Group | Core Treatment Period: Teriflunomide 7 mg | Core Treatment:Teriflunomide 14 mg | Core Treatment: IFN-β-1a | Extended Treatment: Teriflunomide 14 mg (After 7 mg) | Extended Treatment: Teriflunomide 14 mg (After 14 mg) | Extended Treatment: Teriflunomide 14 mg (After IFN-β-1a)
Serious Adverse Events (participants affected / at risk) | 12/110 | 6/110 | 7/101 | 9/90 | 13/88 | 12/59
Other Adverse Events (participants affected / at risk) | 85/110 | 92/110 | 92/101 | 72/90 | 65/88 | 48/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Core Treatment Period: Teriflunomide 7 mg (N=110) | Core Treatment:Teriflunomide 14 mg (N=110) | Core Treatment: IFN-β-1a (N=101) | Extended Treatment: Teriflunomide 14 mg (After 7 mg) (N=90) | Extended Treatment: Teriflunomide 14 mg (After 14 mg) (N=88) | Extended Treatment: Teriflunomide 14 mg (After IFN-β-1a) (N=59)
Appendicitis perforated (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Bacterial pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Tuberculosis (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Cervicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Chronic sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Meningitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Uterine leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haemolysis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hypomania (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Optic neuritis (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Trigeminal neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Eye oedema (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Optic ischaemic neuropathy (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Varicose vein (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Venous stenosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Duodenal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 1
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cervical polyp (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 3 | 1 | 1 | 2 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Core Treatment Period: Teriflunomide 7 mg (N=110) | Core Treatment:Teriflunomide 14 mg (N=110) | Core Treatment: IFN-β-1a (N=101) | Extended Treatment: Teriflunomide 14 mg (After 7 mg) (N=90) | Extended Treatment: Teriflunomide 14 mg (After 14 mg) (N=88) | Extended Treatment: Teriflunomide 14 mg (After IFN-β-1a) (N=59)
Nasopharyngitis (Infections and infestations) | 26 | 24 | 17 | 11 | 9 | 3
Urinary tract infection (Infections and infestations) | 8 | 3 | 6 | 8 | 7 | 3
Bronchitis (Infections and infestations) | 8 | 4 | 2 | 4 | 5 | 4
Upper respiratory tract infection (Infections and infestations) | 8 | 11 | 9 | 2 | 5 | 3
Oral herpes (Infections and infestations) | 9 | 0 | 2 | 1 | 4 | 0
Pharyngitis (Infections and infestations) | 8 | 1 | 3 | 4 | 4 | 5
Influenza (Infections and infestations) | 8 | 9 | 5 | 3 | 2 | 2
Ear infection (Infections and infestations) | 3 | 2 | 2 | 0 | 1 | 3
Gastroenteritis (Infections and infestations) | 5 | 6 | 3 | 7 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 4 | 1 | 2 | 3
Insomnia (Psychiatric disorders) | 7 | 1 | 5 | 2 | 1 | 2
Hypoaesthesia (Nervous system disorders) | 6 | 3 | 2 | 3 | 4 | 3
Dizziness (Nervous system disorders) | 4 | 1 | 6 | 3 | 3 | 0
Headache (Nervous system disorders) | 23 | 17 | 26 | 5 | 3 | 10
Sciatica (Nervous system disorders) | 0 | 0 | 3 | 1 | 3 | 3
Paraesthesia (Nervous system disorders) | 14 | 11 | 8 | 3 | 2 | 3
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 2 | 5 | 6 | 5
Hypertension (Vascular disorders) | 0 | 5 | 4 | 7 | 9 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 4 | 1 | 4 | 2 | 5
Diarrhoea (Gastrointestinal disorders) | 19 | 17 | 9 | 10 | 15 | 8
Abdominal pain (Gastrointestinal disorders) | 5 | 7 | 2 | 6 | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 7 | 7 | 3 | 3 | 3 | 4
Nausea (Gastrointestinal disorders) | 10 | 10 | 4 | 0 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 4 | 4 | 0 | 3 | 1 | 3
Vomiting (Gastrointestinal disorders) | 6 | 9 | 4 | 2 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 22 | 1 | 4 | 1 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 11 | 7 | 5 | 6 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 7 | 4 | 6 | 4 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 7 | 4 | 6 | 3 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 | 5 | 3 | 1 | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 7 | 2 | 1 | 1
Micturition urgency (Renal and urinary disorders) | 2 | 3 | 1 | 2 | 2 | 3
Dysmenorrhoea (Reproductive system and breast disorders) | 3 | 6 | 1 | 1 | 2 | 0
Fatigue (General disorders) | 7 | 6 | 5 | 4 | 4 | 2
Asthenia (General disorders) | 3 | 1 | 9 | 0 | 2 | 3
Pyrexia (General disorders) | 10 | 2 | 3 | 1 | 1 | 0
Influenza like illness (General disorders) | 4 | 4 | 49 | 2 | 0 | 6
Injection site erythema (General disorders) | 0 | 0 | 10 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 12 | 9 | 30 | 5 | 8 | 2
Fall (Injury, poisoning and procedural complications) | 6 | 2 | 2 | 3 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months after trial completion, the Investigator can present or publish results. The investigator provides the sponsor with a copy of the presentation or publication for review and comment at least 30 days in advance of its submission.

The sponsor can delay the submission for a period not exceeding 90 days to allow for filing a patent application or such other measures as sponsor deems appropriate to establish and preserve its proprietary rights.